CLINICAL TRIAL: NCT00034086
Title: Immunologic Consequences of Antiretroviral Therapy Intensification in Subjects With Moderately Advanced HIV-1 Disease: A Follow-Up Study to ACTG 315/375
Brief Title: Study of Anti-HIV Therapy Intensification
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Masking: None | Purpose: Treatment
Other Study IDs: A5136; 10680 (Registry Identifier: DAIDS ES); ACTG A5136; AACTG A5136; ACTG A5140s- Substudy; AACTG A5140s; ACTG A5155s- Substudy; AACTG A5155s
Record Dates: First submitted 2002-04-22; First posted 2002-04-23 (Estimated); Last update posted 2012-05-18 (Estimated); Status verified 2012-05

CONDITIONS: HIV Infections
Keywords: Lopinavir; OspA Protein; HIV-1; HIV Protease Inhibitors; CD4 Lymphocyte Count; Ritonavir; Haemophilus Vaccines; HAART; Pneumococcal Vaccines; tenofovir disoproxil
MeSH Terms: conditions — HIV Infections | interventions — Lopinavir; lamivudine, zidovudine drug combination; Tenofovir; Pneumococcal Vaccines; Lamivudine; Stavudine; Zidovudine; Didanosine; OspA protein; HibTITER protein, Haemophilus influenzae

INTERVENTIONS:
Drug: Lopinavir/Ritonavir
Drug: Lamivudine/Zidovudine
Drug: Tenofovir disoproxil fumarate
Biological: Pneumococcal Vaccine, Polyvalent (23-valent)
Drug: Lamivudine
Drug: Stavudine
Drug: Zidovudine
Drug: Didanosine
Biological: Lyme Disease Vaccine Recombinant OspA
Biological: Haemophilus B Conjugate Vaccine

SUMMARY:
The purpose of this study is to see how the body's immune system changes after replacing and adding new anti-HIV drugs to a patient's current anti-HIV therapy. This study will also see whether adding drugs is safe. Patients who take part in A5136 are also eligible to take part in 2 substudies. The purpose of substudy A5140s is to see how many latently infected cells (cells in which the HIV virus survives) are in the lymph node (small, rounded structures that make disease-fighting cells). Substudy A5155s will be performed to see how many latently infected cells are in the blood before and after replacing and adding anti-HIV drugs.

ACTG A5136 is a follow-up study to ACTG 315 and ACTG 375, which were designed to examine the effects of highly active antiretroviral therapy (HAART) in certain HIV-infected patients. Many HIV-infected patients have undergone long-term anti-HIV therapy and have had the virus suppressed. However, most of these patients still have problems with their immune systems. The reason for these problems is unknown. This study may help researchers understand what causes immune system problems in people who have low levels of HIV in their blood.

DETAILED DESCRIPTION:
ACTG 315 and its follow-up study, ACTG 375, were designed to examine the immunologic and virologic consequences of highly active antiretroviral therapy (HAART) in patients with moderately advanced HIV-1 disease. At the conclusion of ACTG 375, patients eligible for participation in ACTG A5136 will have received over 5 years of antiretroviral therapy. Despite long-term therapy and long-term maximal viral suppression in most patients, significant immune defects such as impaired response to antigens, including HIV, abnormally low CD4 cell counts, abnormally high immune activation, and decreased expression of CD28 persist. It is uncertain whether these defects persist as a result of irreversible damage inflicted by HIV infection or ongoing immune perturbation resulting from continuous low-level HIV replication. Cellular reservoirs of HIV that persist (despite undetectable plasma viral load) may contribute to persistent immune activation and impaired immune function. A great deal of information on the relationship between low-level viral replication and persistent immune impairment may be gained by investigating these patients before and after intensification of their antiretroviral therapy regimens.

Patients continue to receive their ACTG 375 antiretroviral therapy until they register to A5136. Following entry evaluations, patients replace the protease inhibitors (PIs) in their ACTG 375 regimen with lopinavir/ritonavir (LPV/r), add tenofovir disoproxil fumarate (TDF) to their regimen, and maintain the rest of their ACTG 375 regimen for 48 weeks. Patients have clinic visits at entry and at Weeks 4, 12, and 16. After 24 weeks, patients have clinic visits every 12 weeks. Blood is drawn at these visits for viral load, immune response, and other routine tests. A skin test, a urine sample collection, and a pregnancy test (for women of reproductive potential) are also performed at entry. Patients also receive immunizations. At Weeks 12 and 16, a lyme vaccine, polyvalent is administered. At Week 36, lyme vaccine, polyvalent; pneumococcal vaccine, polyvalent; and haemophilus b conjugate (HIB) vaccine are administered [AS PER AMENDMENT 05/14/02: Lyme disease vaccine has been removed from the study due to unavailability]. At Week 48, skin tests are performed. Week 52 is the final clinic visit, at which blood is drawn and a urine sample is taken.

Patients who participate in substudy A5140s undergo 2 lymph node aspirates, at entry and at Week 48. Patients participating in substudy A5155s have blood drawn at screening and Week 48.

ELIGIBILITY:
Inclusion Criteria

Patients may be eligible for this study if they:

* Have completed ACTG 375 within 2 weeks of finishing Week 230.
* Have a viral load less than 400 copies/ml within 90 days prior to study entry.
* Agree not to become pregnant or to impregnate during the study. The female patient/male partner must use acceptable methods of contraception while receiving study drugs and for 1 month after stopping the drugs. Women and men who cannot have children are eligible without requiring the use of contraception, but they must provide acceptable documentation of menopause, sterilization, or lack of sperm cells.

Exclusion Criteria

Patients may not be eligible for this study if they:

* Need to use certain drugs within 30 days of study entry.
* Have taken any immunomodulatory therapies within 30 days prior to study entry unless approved by the protocol chairs.
* Have a history of serious kidney problems.
* Are allergic or sensitive to the study drugs.
* Are pregnant or breast-feeding.
* Have an alcohol or drug dependency that, in the opinion of the investigator, would interfere with the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 22
Dates: Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Smith, Study Chair; Hernan Valdez, Study Chair
Locations (3):
- United States (3):
  - University of Colorado Hospital CRS, Aurora, Colorado
  - Rush Univ. Med. Ctr. ACTG CRS, Chicago, Illinois
  - Case CRS, Cleveland, Ohio